CLINICAL TRIAL: NCT02655328
Title: Diagnosis et Treatment of Asthma in Athlete : Boundary Between Disease and Doping
Acronym: SALBEXO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08 301 03
Record Dates: First submitted 2015-07-10; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
Keywords: asthma; athlete
MeSH Terms: conditions — Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- athlete under asthma treatment (Experimental): athlete suffering from asthma blood sample urine sample
  Interventions: Other: blood sample; Other: urine sample

INTERVENTIONS:
Other: blood sample — blood sample
Other: urine sample — urine sample

SUMMARY:
This study will determine the pharmacokinetic profile of the salbutamol concentration in the urine while athletes are resting or during exercise.

ELIGIBILITY:
Inclusion Criteria:

* patient who hold a license in a sport federation, and do at least 8 hours of sport each week
* asthmatic patient

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
impact of exercise on pharmacokinetics profile | 4 days
  impact of exercise on pharmacokinetics profile of salbutamol concentration in urine

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rivière, MD, Principal Investigator — UH Toulouse
Locations (1):
- UH Toulouse, Toulouse, France